CLINICAL TRIAL: NCT03869346
Title: Impact of CYP3A4*1G Polymorphism on Non-analgesic Effects of Fentanyl in Chinese Han Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Principal Investigator, Yanqi, Attending, Peking University People's Hospital
Other Study IDs: NAOOP
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Fentanyl

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 200 blood samples were withdrawn
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- GG: wild-type homozygote (CYP3A4*1/*1, GG)
- GA: mutant heterozygote (CYP3A4*1/*1G, GA),
- AA: mutant homozygote (CYP3A4*1G/*1G, AA)

SUMMARY:
Purpose: This study aimed to investigate the impact of CYP3A4*1G genetic polymorphism on non-analgesic effects of fentanyl in Chinese Han patients. Methods: 200 patients receiving elective surgery under general anesthesia were recruited into this study. Venous blood was withdrawn for genotyping of CYP3A4*1G before operation. Fentanyl 2 µg/kg was administered preoperatively. Bispectral Index (BIS), Respiratory rate(RR), etc at Tb (entering room), T0 (drug administration), T1 (2min), T2 (4min), T3(6min), T4(8min), T5(10min), T6(20min) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists GradeⅠ-II,Patients undergo elective surgery for benign Reproductive diseases (including laparoscopic ovarian cyst removal, laparoscopic tubal ligation, laparoscopic tubal drainage, laparoscopic salpingoplasty, etc.) or breast disease.
* Aged 18-45 years
* Body Mass Index 18-25kg/m2,body weight 40-65 kilograms
* Agreed to participate the research

Exclusion Criteria:

* Difficult airway
* upper respiratory tract infection within 2 weeks
* history of allergy or long-term use of propofol and opioids
* self-rating anxiety scale before operation indicates anxiety
* pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 Chinese Han patients receiving elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-10 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
bispectral index | 20 min after administration
  bispectral index(BIS): assessing the sedation, placed on the patient's forehead, BIS values 0-100, and the higher score means patients are more conscious
respiratory rate | 20 min after administration
  Number of breaths per minute
CYP3A4*1G Polymorphism | 1 week after operation
  The patients were classified by genotype including wild-type homozygote (CYP3A4*1/*1, GG), mutant heterozygote (CYP3A4*1/*1G, GA), and mutant homozygote (CYP3A4*1G/*1G, AA).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, Professor, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No